CLINICAL TRIAL: NCT01388634
Title: Nationwide Analysis of Prolonged Hospital Stay and Readmission After Elective Ventral Hernia Repair
Brief Title: Prolonged Hospital Stay and Readmission After Elective Ventral Hernia Repair
Acronym: LOSHERNIA
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, Zealand University Hospital
Other Study IDs: Køge hospital
Record Dates: First submitted 2011-06-27; First posted 2011-07-06 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Ventral Hernia
Keywords: Length of hospital stay; readmission; ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study cohort: Patients with prolonged length of hospital stay (>5 days) or readmission after ventral hernia repair
- control group: Patients without prolonged length of hospital stay (>5 days) or readmission after ventral hernia repair

SUMMARY:
The aim of the present study was to analyse factors associated with prolonged length of hospital stay, readmission and death in a nationwide group of patients undergoing elective ventral hernia repair in search for areas of interest to improve outcome after ventral hernia surgery

DETAILED DESCRIPTION:
Detailed analysis of reasons for prolonged hospital stay and readmission in patients undergoing a ventral hernia repair

ELIGIBILITY:
Inclusion Criteria:

* patients with elective ventral hernia repair in Denmark 2008

Exclusion Criteria:

* emergency repairs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients registered in The Danish Ventral Hernia Database in 2008
Sampling Method: Non-Probability Sample
Enrollment: 2258 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 1 week
  analyse factors associated with prolonged length of hospital stay (minimum 5 days).

SECONDARY OUTCOMES:
Readmission | 30 days
  reasons for readmission after a ventral hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Helgstrand, MD, Principal Investigator — Dept. surgery Køge hospital
Locations (1):
- Dept. of surgery, Køge Hospital, Køge, Denmark

REFERENCES:
- [Derived] Helgstrand F, Rosenberg J, Kehlet H, Bisgaard T. Nationwide analysis of prolonged hospital stay and readmission after elective ventral hernia repair. Dan Med Bull. 2011 Oct;58(10):A4322. PMID 21975153